CLINICAL TRIAL: NCT01459016
Title: An Exploratory Study of Brain Imaging Biomarkers in Patients With Alzheimer's Pathology Receiving Standard of Care
Brief Title: A Non-drug Methods Study in Participants With Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 14162; I4O-MC-BACH (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-10-12; First posted 2011-10-25 (Estimated); Results first posted 2017-02-13 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-05

CONDITIONS: Alzheimer's Disease
Keywords: Mild Cognitive Impairment; Brain Imaging Biomarkers; Magnetic resonance imaging biomarker; Positron Emission Tomography
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Imaging Biomarkers (Experimental)
  Interventions: Other: PET scan using florbetapir; Other: MRI Scan

INTERVENTIONS:
Other: PET scan using florbetapir — A single intravenous microdose of 260 MBq (7 mCi) 18F-AV-45 (florbetapir F 18) will be administered.
  Other Names: AV-45
Other: MRI Scan — Three different measurements will be taken: volumetric MRI (vMRI), diffusion tensor imaging (DTI), and resting state functional MRI (rsfMRI). In addition, radiological MRI scans will be taken to monitor vasogenic edema and microhemorrhages.

SUMMARY:
This study will investigate the volume, function and composition of the brain using magnetic resonance imaging (MRI) and positron emission tomography (PET) scanning technology in participants with memory complaints or early signs of Alzheimer's pathology.

DETAILED DESCRIPTION:
After trial initiation, the protocol was amended to extend the single observation time period (6 to 9 months) to two time points (6 and 12 months), and to focus on prodromal AD (Mini-Mental State Examination [MMSE] 23-30 inclusive, Free and Cued Selective Reminding Test [FCSRT] less than or equal to [≤] 24 for free recall or ≤ 44 for total recall). Participants enrolled under the original protocol were allowed to continue in the extension study if they so desired, and if they met the new inclusion criteria. Due to the number of participants that completed the extended trial, no sub-group analysis was performed based on which amendment the participants entered under.

ELIGIBILITY:
Inclusion Criteria:

* Present with prodromal Alzheimer's Disease (AD) or mild AD based on the disease diagnostic criteria
* Are men or post-menopausal women, at least 55 years of age. Post-menopausal women are defined as women who have had a hysterectomy and/or bilateral oophorectomy; or who have been amenorrheic for at least 2 years
* Have a caretaker/study informant who provides a separate written informed consent to participate. If a caretaker/study informant cannot continue, one replacement is allowed
* Gradual and progressive change in memory function reported by participants or informants over more than 6 months
* Objective evidence of significantly impaired episodic memory characteristic of hippocampal dysfunction on testing: Free and Cued Selective Reminding Test (FCSRT): less than or equal to (≤) 16 for free recall or ≤ 40 for total recall. Protocol amendment: FCSRT ≤ 24 for free recall or ≤ 44 for total recall
* Clinical Dementia Rating (CDR) equals 0.5 or 1, Memory box score greater than or equal to 0.5
* Mini Mental Scale Examination (MMSE) 20-30. Protocol amendment: MMSE 23-30, inclusive
* Positive florbetapir F 18 scan
* Participants must meet all of the Disease Diagnostic Criteria to be considered for enrollment

Exclusion Criteria:

* Diagnosis or history of other possible etiology of dementia, including but not limited to other neurodegenerative disorders
* Frontotemporal dementia, Lewy body disease, vascular dementia, Huntington's Disease or concomitant Parkinson's disease, progressive supranuclear palsy (PSNP) or other movement disorder
* Has B12 <200 pg/L or folate <7.5 nmol/L indicating vitamin deficiency
* Has a history within the past 5 years of a serious infectious disease affecting the brain, including meningitis, or encephalitis
* Significant history of alcoholism or substance abuse (at the judgment of the investigator)
* Severe or recurrent head injury that is clinically relevant to the disease under study, (that is, with permanent neurological/cognitive sequelae)
* Onset of dementia following heart surgery or cardiac arrest
* Diagnosis or history of cerebrovascular disease (for example, stroke, transient ischemic attack), severe carotid stenosis, cerebral hemorrhage, intracranial tumor, subarachnoid hemorrhage, or subdural hematoma that could contribute to the subject's current cognitive or functional status, impair ability to fully participate in the trial or that may impact status
* Has had a Positron Emission Tomography (PET) within 6 months of the scheduled imaging follow-up
* Greater than 4 cerebral microhemorrhages (CMH) on T2* -weighted gradient-recalled echo sequences (regardless of their anatomical or diagnostic characterization as "possible" or "definite"), a single area of superficial siderosis, or prior evidence of macrohemorrhage
* Any indications of severe deep white matter lesions or vasogenic edema that present as hyperintense regions on the Fluid Attenuated Inversion Recovery (FLAIR) sequence, or other clinically relevant findings observed on the Magnetic Resonance Imaging (MRI) scans
* Specific exclusionary brain MRI findings, as determined by the investigator in consultation with the sponsor, that could either contribute to the participant's current cognitive or functional decline impair ability to fully participate in the trial or that may impact status during the trial (for example, brain tumors or other non-vascular structural abnormalities like hydrocephalus)
* History within the past 5 years of a primary or recurrent malignant disease with the exception of resected cutaneous squamous cell carcinoma in situ, basal cell carcinoma, cervical carcinoma in situ, or in situ prostate cancer with a normal prostate-specific antigen (PSA) post resection
* History of clinically significant cardiovascular or renal events
* Diastolic blood pressure of 95 or more and systolic blood pressure of 160 or more in sitting position after at least 5 minutes of rest
* Any history of seizure
* History of clinically significant head trauma or clinically significant unexplained loss of consciousness within the last 5 years (as determined by the investigator in consultation with the Sponsor)
* A current Axis I diagnosis of major depressive disorder or other psychiatric illness (Diagnostic and Statistical Manual Revised Fourth Edition [DSM-IV-TR]) criteria per the investigator's judgment. (Note: Participants on a stable antidepressant and/or anxiolytic treatment may participate.)
* Having suicidal ideations, or attempted suicide in the past 15 years
* History of schizophrenia, bipolar disorder, or other severe mental illness
* Known history of alcohol or drug abuse (as defined by the DSM-IV-TR) within 5 years prior to enrolling or a positive result regarding use of illicit drugs on the drug screening test
* Chronic hepatic diseases as indicated by liver function test abnormalities (alanine trasaminase [ALT], aspartate transaminase [AST], bilirubin, or gamma-glutamyl transferase [GGT] above 2 times upper limit of normal), positive serology for Hepatitis B or C, or other manifestations of liver disease
* Has compromised renal function at screening, as determined by creatinine clearance <30 mL/min based on Cockcroft-Gault calculation of creatinine clearance
* History of asthma, chronic obstructive pulmonary disease, or other chronic respiratory conditions
* Known positive human immunodeficiency virus (HIV) status, history of syphilitic infection
* A clinically significant abnormality in the 12-lead electrocardiograms (ECG), including complete heart block, bradycardia (heart rate <50 beats/minute), tachycardia (heart rate ≥95 beats/minute), sinus pauses >2 seconds, second or third degree heart block, QTc >450 msec for males or QTc >470 for females
* Treatment with an investigational small molecule within 1 year preceding the first study period, or participation in a trial with active or passive immunization against amyloid if participant was assigned to the active treatment arm
* Fulfillment of any contraindications to a 3T magnetic resonance imaging (MRI) scan (for example, subjects with non-removable ferromagnetic implants (such as cardiac pacemaker), aneurysm clips or other foreign bodies, or subjects with claustrophobic symptoms that would contraindicate an MRI scan)
* Sensitivity to florbetapir F 18
* Are not capable of swallowing whole oral medications
* Abnormal thyroid function

  * Thyroid stimulating hormone (TSH) values are outside of the normal range 0.3-5.6 mIU/L. (NOTE: Participants with stable treatment of hypothyroidism and with normal value of TSH will be allowed to enter the study)

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2011-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri, 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (16):
- France (16):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cahors
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Castres
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Foix
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lavaur
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Léon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Limoges
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marseille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montauban
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nancy
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rennes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Strasbourg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toulouse
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tours
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vic-en-Bigorre

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care: Participants with prodromal to mild Alzheimer's Disease (AD) underwent a florbetapir F 18 positron emission tomography (PET) scan. (Single intravenous microdose of 260 to 370 megabecquerels (MBq) [7 to 10 millicuries (mCi)] of florbetapir.) Those who tested amyloid positive and met other entry criteria received standard of care for up to 12 months (mos). No therapeutic investigational drug intended to treat AD was administered.
Period: Overall Study
Arm/Group | Standard of Care
Started | 56
Completed | 41
Not Completed | 15
Not completed — Withdrawal by Subject | 11
Not completed — Amendment Discontinuation Criteria | 4

BASELINE CHARACTERISTICS:
Population: All participants who enrolled in the study.
Groups:
- Standard of Care: Participants with prodromal to mild AD underwent a florbetapir F 18 PET scan. (Single intravenous microdose of 260 to 370 MBq [7 to 10 mCi] of florbetapir.) Those who tested amyloid positive and met other disease diagnostic criteria received standard of care for up to 12 mos. No therapeutic investigational drug intended to treat AD was administered.
Arm/Group | Standard of Care
Number analyzed (Participants) | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.2 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 34
Region of Enrollment [Count of Participants; unit: Participants]
  France | 56

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Volumetric Magnetic Resonance Imaging (vMRI) - Brain Boundary Shift Integral (BBSI) and Ventricular Boundary Shift Integral (VBSI)
Description: BBSI and VBSI were calculated based on the voxel-wise difference between co-registered baseline and follow-up scans. Least squares (LS) mean value was controlled for baseline value and visit.
Time Frame: Baseline, 6 Mos; Baseline, 12 Mos
Population: All participants who enrolled in the study and had an evaluable MRI at the designated time point.
Measure: Least Squares Mean (95% Confidence Interval); unit: milliliters (mL)
Arm/Group | Standard of Care
Number analyzed (Participants) | 56
milliliters (mL)
  BBSI - 6 Mos: number analyzed (Participants) | 43
  BBSI - 6 Mos | 6.349 [3.735 to 8.963]
  BBSI - 12 Mos: number analyzed (Participants) | 31
  BBSI - 12 Mos | 11.663 [8.608 to 14.719]
  VBSI - 6 Mos: number analyzed (Participants) | 45
  VBSI - 6 Mos | 2.016 [1.361 to 2.671]
  VBSI - 12 Mos: number analyzed (Participants) | 31
  VBSI - 12 Mos | 4.196 [3.088 to 5.303]

2. Primary Outcome: Change From Baseline in Volumetric Magnetic Resonance Imaging (vMRI) - Hippocampus Volume Average Percent (%) Change (Chg)
Description: Automated hippocampal volumetry was performed using the Learning Embeddings for Atlas Propagation (LEAP) algorithm. LS mean value was controlled for baseline value and visit.
Time Frame: Baseline, 6 Mos; Baseline, 12 Mos
Population: All participants who enrolled in the study and had an evaluable MRI at the designated time point.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of hippocampus volume average
Arm/Group | Standard of Care
Number analyzed (Participants) | 56
percentage of hippocampus volume average
  Hippocampus Volume Average % Chg - 6 Mos: number analyzed (Participants) | 44
  Hippocampus Volume Average % Chg - 6 Mos | -1.693 [-2.273 to -1.113]
  Hippocampus Volume Average % Chg - 12 Mos: number analyzed (Participants) | 30
  Hippocampus Volume Average % Chg - 12 Mos | -3.057 [-3.884 to -2.231]

3. Primary Outcome: Change From Baseline in Resting State Functional Magnetic Resonance Imaging (rsfMRI)
Description: Distributed functional connectivity in selected brain networks was calculated from the rsfMRI scans. Values were derived from low-frequency (0.01-0.1 hertz [Hz]) temporal correlations between different regions over the approximately 6-minute rsfMRI time series scan. Distributed measures of functional connectivity were calculated as the mean Pearson correlation between the average low-frequency time courses in predefined sets of regions of interest (ROI) within the default mode network (DMN), salience network (SN) and sensorimotor networks (SMN). LS mean value was controlled for baseline value and visit.
Time Frame: Baseline, 6 Mos; Baseline, 12 Mos
Population: All participants who enrolled in the study and had an evaluable MRI at the designated time point.
Measure: Least Squares Mean (95% Confidence Interval); unit: arbitrary units (au)
Arm/Group | Standard of Care
Number analyzed (Participants) | 56
arbitrary units (au)
  Anterior DMN - 6 Mos: number analyzed (Participants) | 41
  Anterior DMN - 6 Mos | 0.017 [-0.033 to 0.067]
  Anterior DMN - 12 Mos: number analyzed (Participants) | 28
  Anterior DMN - 12 Mos | 0.031 [-0.017 to 0.080]
  Anterior SN - 6 Mos: number analyzed (Participants) | 41
  Anterior SN - 6 Mos | -0.012 [-0.043 to 0.019]
  Anterior SN -12 Mos: number analyzed (Participants) | 28
  Anterior SN -12 Mos | -0.025 [-0.065 to 0.014]
  DMN - 6 Mos: number analyzed (Participants) | 41
  DMN - 6 Mos | -0.029 [-0.060 to 0.001]
  DMN - 12 Mos: number analyzed (Participants) | 28
  DMN - 12 Mos | -0.031 [-0.061 to -0.001]
  Posterior DMN - 6 Mos: number analyzed (Participants) | 41
  Posterior DMN - 6 Mos | -0.061 [-0.120 to -0.002]
  Posterior DMN - 12 Mos: number analyzed (Participants) | 28
  Posterior DMN - 12 Mos | -0.058 [-0.096 to -0.021]
  Posterior SN - 6 Mos: number analyzed (Participants) | 41
  Posterior SN - 6 Mos | -0.012 [-0.045 to 0.021]
  Posterior SN - 12 Mos: number analyzed (Participants) | 28
  Posterior SN - 12 Mos | 0.001 [-0.040 to 0.043]
  SN - 6 Mos: number analyzed (Participants) | 41
  SN - 6 Mos | -0.021 [-0.048 to 0.005]
  SN - 12 Mos: number analyzed (Participants) | 28
  SN - 12 Mos | -0.008 [-0.043 to 0.027]
  SMN - 6 Mos: number analyzed (Participants) | 41
  SMN - 6 Mos | 0.041 [0.009 to 0.072]
  SMN - 12 Mos: number analyzed (Participants) | 28
  SMN - 12 Mos | -0.013 [-0.060 to 0.034]

4. Primary Outcome: Change From Baseline in Diffusion Tensor Imaging (DTI) Using Fractional Anisotropy (FA)
Description: DTI scans used FA to measure water diffusion directionality in selected white matter (WM) tracts. ROI: Corpus collosum (CC), internal capsule (IC), posterior cingulum bundle (PCB), temporal white matter (TWM), uncinate fasciculus (UF), superior longitudinal fasciculus (SLF). LS mean value was controlled for baseline value and visit.
Time Frame: Baseline, 6 Mos; Baseline, 12 Mos
Population: All participants who enrolled in the study and had an evaluable MRI at the designated time point.
Measure: Least Squares Mean (95% Confidence Interval); unit: au
Arm/Group | Standard of Care
Number analyzed (Participants) | 56
au
  Mean FA, CC (Genu) - 6 Mos: number analyzed (Participants) | 44
  Mean FA, CC (Genu) - 6 Mos | -0.024 [-0.046 to -0.003]
  Mean FA, CC (Genu) - 12 Mos: number analyzed (Participants) | 30
  Mean FA, CC (Genu) - 12 Mos | -0.021 [-0.041 to -0.001]
  Mean FA, CC (Splenium) - 6 Mos: number analyzed (Participants) | 44
  Mean FA, CC (Splenium) - 6 Mos | -0.016 [-0.043 to 0.012]
  Mean FA, CC (Splenium) - 12 Mos: number analyzed (Participants) | 30
  Mean FA, CC (Splenium) - 12 Mos | 0.009 [-0.026 to 0.043]
  Mean FA, IC (Left) - 6 Mos: number analyzed (Participants) | 44
  Mean FA, IC (Left) - 6 Mos | -0.043 [-0.066 to -0.020]
  Mean FA, IC (Left) - 12 Mos: number analyzed (Participants) | 30
  Mean FA, IC (Left) - 12 Mos | -0.020 [-0.043 to 0.003]
  Mean FA, IC (Right) - 6 Mos: number analyzed (Participants) | 44
  Mean FA, IC (Right) - 6 Mos | -0.046 [-0.067 to -0.025]
  Mean FA, IC (Right) - 12 Mos: number analyzed (Participants) | 30
  Mean FA, IC (Right) - 12 Mos | -0.020 [-0.038 to -0.002]
  Mean FA, PCB (Left) - 6 Mos: number analyzed (Participants) | 44
  Mean FA, PCB (Left) - 6 Mos | 0.000 [-0.012 to 0.013]
  Mean FA, PCB (Left) - 12 Mos: number analyzed (Participants) | 30
  Mean FA, PCB (Left) - 12 Mos | 0.010 [0.003 to 0.017]
  Mean FA, PCB (Right) - 6 Mos: number analyzed (Participants) | 44
  Mean FA, PCB (Right) - 6 Mos | 0.010 [-0.001 to 0.021]
  Mean FA, PCB (Right) - 12 Mos: number analyzed (Participants) | 30
  Mean FA, PCB (Right) - 12 Mos | 0.003 [-0.008 to 0.015]
  Mean FA, TWM (Left) - 6 Mos: number analyzed (Participants) | 44
  Mean FA, TWM (Left) - 6 Mos | -0.017 [-0.028 to -0.006]
  Mean FA, TWM (Left) - 12 Mos: number analyzed (Participants) | 30
  Mean FA, TWM (Left) - 12 Mos | -0.011 [-0.022 to 0.000]
  Mean FA, TWM (Right) - 6 Mos: number analyzed (Participants) | 44
  Mean FA, TWM (Right) - 6 Mos | -0.014 [-0.022 to -0.005]
  Mean FA, TWM (Right) - 12 Mos: number analyzed (Participants) | 30
  Mean FA, TWM (Right) - 12 Mos | -0.009 [-0.019 to 0.001]
  Mean FA, UF (Left) - 6 Mos: number analyzed (Participants) | 44
  Mean FA, UF (Left) - 6 Mos | -0.027 [-0.045 to -0.010]
  Mean FA, UF (Left) - 12 Mos: number analyzed (Participants) | 30
  Mean FA, UF (Left) - 12 Mos | 0.010 [-0.007 to 0.027]
  Mean FA, UF (Right) - 6 Mos: number analyzed (Participants) | 44
  Mean FA, UF (Right) - 6 Mos | -0.032 [-0.049 to -0.015]
  Mean FA, UF (Right) - 12 Mos: number analyzed (Participants) | 30
  Mean FA, UF (Right) - 12 Mos | 0.005 [-0.009 to 0.020]
  Mean FA, SLF (Left) - 6 Mos: number analyzed (Participants) | 44
  Mean FA, SLF (Left) - 6 Mos | -0.014 [-0.025 to -0.003]
  Mean FA, SLF (Left) - 12 Mos: number analyzed (Participants) | 30
  Mean FA, SLF (Left) - 12 Mos | -0.003 [-0.014 to 0.007]
  Mean FA, SLF (Right) - 6 Mos: number analyzed (Participants) | 44
  Mean FA, SLF (Right) - 6 Mos | -0.006 [-0.019 to 0.007]
  Mean FA, SLF (Right) - 12 Mos: number analyzed (Participants) | 30
  Mean FA, SLF (Right) - 12 Mos | 0.002 [-0.009 to 0.012]

5. Primary Outcome: Change From Baseline in Diffusion Tensor Imaging (DTI) Using Mean Diffusivity (MD)
Description: DTI scans used MD to measure the overall magnitude of water diffusion in selected WM tracts, without specific regard to directionality. ROI: CC, IC, PCB, TWM, UF, SLF. LS mean value was controlled for baseline value and visit.
Time Frame: Baseline, 6 Mos; Baseline, 12 Mos
Population: All participants who enrolled in the study and had an evaluable MRI at the designated time point.
Measure: Least Squares Mean (95% Confidence Interval); unit: square meters per second (m²/sec) * 10¹⁰
Arm/Group | Standard of Care
Number analyzed (Participants) | 56
square meters per second (m²/sec) * 10¹⁰
  Mean MD, CC (Genu) - 6 Mos: number analyzed (Participants) | 44
  Mean MD, CC (Genu) - 6 Mos | 0.201 [-0.157 to 0.559]
  Mean MD, CC (Genu) - 12 Mos: number analyzed (Participants) | 30
  Mean MD, CC (Genu) - 12 Mos | 0.761 [-0.280 to 1.802]
  Mean MD, CC (Splenium) - 6 Mos: number analyzed (Participants) | 44
  Mean MD, CC (Splenium) - 6 Mos | 0.663 [-0.114 to 1.440]
  Mean MD, CC (Splenium) - 12 Mos: number analyzed (Participants) | 30
  Mean MD, CC (Splenium) - 12 Mos | -0.519 [-0.956 to -0.082]
  Mean MD, IC (Left) - 6 Mos: number analyzed (Participants) | 44
  Mean MD, IC (Left) - 6 Mos | 0.410 [0.043 to 0.777]
  Mean MD, IC (Left) - 12 Mos: number analyzed (Participants) | 30
  Mean MD, IC (Left) - 12 Mos | 0.164 [-0.107 to 0.435]
  Mean MD, IC (Right) - 6 Mos: number analyzed (Participants) | 44
  Mean MD, IC (Right) - 6 Mos | 0.441 [0.203 to 0.679]
  Mean MD, IC (Right) - 12 Mos: number analyzed (Participants) | 30
  Mean MD, IC (Right) - 12 Mos | 0.280 [0.120 to 0.440]
  Mean MD, PCB (Left) - 6 Mos: number analyzed (Participants) | 44
  Mean MD, PCB (Left) - 6 Mos | -0.062 [-0.326 to 0.203]
  Mean MD, PCB (Left) - 12 Mos: number analyzed (Participants) | 30
  Mean MD, PCB (Left) - 12 Mos | 0.175 [-0.087 to 0.436]
  Mean MD, PCB (Right) - 6 Mos: number analyzed (Participants) | 44
  Mean MD, PCB (Right) - 6 Mos | 0.114 [-0.156 to 0.385]
  Mean MD, PCB (Right) - 12 Mos: number analyzed (Participants) | 30
  Mean MD, PCB (Right) - 12 Mos | 0.297 [0.053 to 0.541]
  Mean MD TWM (Left) - 6 Mos: number analyzed (Participants) | 44
  Mean MD TWM (Left) - 6 Mos | -0.014 [-0.280 to 0.251]
  Mean MD TWM (Left) - 12 Mos: number analyzed (Participants) | 30
  Mean MD TWM (Left) - 12 Mos | -0.010 [-0.295 to 0.274]
  Mean MD TWM (Right) - 6 Mos: number analyzed (Participants) | 44
  Mean MD TWM (Right) - 6 Mos | 0.243 [-0.047 to 0.533]
  Mean MD TWM (Right) - 12 Mos: number analyzed (Participants) | 30
  Mean MD TWM (Right) - 12 Mos | 0.285 [0.077 to 0.493]
  Mean MD, UF (Left) - 6 Mos: number analyzed (Participants) | 44
  Mean MD, UF (Left) - 6 Mos | -0.150 [-0.518 to 0.218]
  Mean MD, UF (Left) - 12 Mos: number analyzed (Participants) | 30
  Mean MD, UF (Left) - 12 Mos | -0.600 [-1.005 to -0.196]
  Mean MD, UF (Right) - 6 Mos: number analyzed (Participants) | 44
  Mean MD, UF (Right) - 6 Mos | 0.240 [-0.200 to 0.681]
  Mean MD, UF (Right) - 12 Mos: number analyzed (Participants) | 30
  Mean MD, UF (Right) - 12 Mos | -0.289 [-0.649 to 0.072]
  Mean MD SLF (Left) - 6 Mos: number analyzed (Participants) | 44
  Mean MD SLF (Left) - 6 Mos | 0.083 [-0.070 to 0.237]
  Mean MD SLF (Left) - 12 Mos: number analyzed (Participants) | 30
  Mean MD SLF (Left) - 12 Mos | -0.007 [-0.108 to 0.094]
  Mean MD SLF (Right) - 6 Mos: number analyzed (Participants) | 44
  Mean MD SLF (Right) - 6 Mos | 0.085 [-0.113 to 0.284]
  Mean MD SLF (Right) - 12 Mos: number analyzed (Participants) | 30
  Mean MD SLF (Right) - 12 Mos | 0.097 [-0.004 to 0.197]

6. Secondary Outcome: Baseline Brain Amyloid Load Using Positron Emission Tomography (PET) and Florbetapir
Description: Composite summary standardized uptake value ratio (SUVR) normalized to mean whole cerebellum. Regions used for composite summary were posterior cingulum, anterior cingulum, parietal cortex, lateral temporal cortex and frontal cortex.
Time Frame: Baseline
Population: All participants with an amyloid positive florbetapir F 18 PET scan at baseline.
Measure: Mean (Standard Deviation); unit: SUVR unit 1
Arm/Group | Standard of Care
Number analyzed (Participants) | 56
SUVR unit 1 | 1.581 (0.200)

7. Secondary Outcome: Number of Participants With Vasogenic Edema on MRI Scan at a Field Strength of 3 Tesla (3T)
Time Frame: Baseline
Population: All participants who had an MRI during screening and were classified as screen failures.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care
Number analyzed (Participants) | 42
Participants | 4

8. Secondary Outcome: Number of Participants With Microhemorrhage on MRI Scan at a Field Strength of 3T
Time Frame: Baseline, 6 Mos; Baseline, 12 Mos
Population: All participants who enrolled in the study and had an evaluable MRI at the designated time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care
Number analyzed (Participants) | 56
Participants
  Baseline | 16
  6 Mos: number analyzed (Participants) | 46
  6 Mos | 12
  12 Mos: number analyzed (Participants) | 31
  12 Mos | 9

9. Secondary Outcome: Change From Baseline in the Mini Mental State Examination (MMSE) Total Score
Description: The MMSE is a brief screening instrument used to assess cognitive function (orientation, memory, attention, ability to name objects, follow verbal/written commands, write a sentence, and copy figures). Total score ranges from 0 to 30; lower score indicates greater disease severity. LS mean value was controlled for baseline value and visit.
Time Frame: Baseline, 6 Mos; Baseline, 12 Mos
Population: All participants who enrolled in the study and completed the scale at the designated time point.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Standard of Care
Number analyzed (Participants) | 56
units on a scale
  6 Mos: number analyzed (Participants) | 48
  6 Mos | -1.2 [-2.0 to -0.5]
  12 Mos: number analyzed (Participants) | 32
  12 Mos | -1.8 [-2.7 to -0.8]

10. Secondary Outcome: Change From Baseline in the Alzheimer's Disease Assessment Scale Extended Cognitive Subscale (ADAS-Cog14) Total Score
Description: The ADAS-Cog14 is the ADAS-Cog11 augmented with delayed free recall, digit cancellation, and maze completion measures. A score of 0 to 10 for delayed free recall and a conversion code of 0 to 5 for digit cancellation and maze completion provide total score ranges for this extended ADAS-Cog14 of 0 to 90. Higher scores indicate greater disease severity. LS mean value was controlled for baseline value and visit.
Time Frame: Baseline, 6 Mos; Baseline, 12 Mos
Population: All participants who enrolled in the study and completed the scale at the designated time point.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Standard of Care
Number analyzed (Participants) | 56
units on a scale
  6 Mos: number analyzed (Participants) | 46
  6 Mos | 0.1 [-1.6 to 1.8]
  12 Mos: number analyzed (Participants) | 31
  12 Mos | 0.7 [-1.7 to 3.1]

11. Secondary Outcome: Change From Baseline in the Clinical Dementia Rating (CDR) Total Score
Description: The CDR is a semi-structured interview of participants and their caregivers. Participant's cognitive status is rated across 6 domains of functioning, including memory, orientation, judgment/problem solving, community affairs, home/hobbies, and personal care. Severity score assigned for each of 6 domains; Total score ranges from 0 to 18. Higher scores indicate greater disease severity. LS mean value was controlled for baseline value and visit.
Time Frame: Baseline, 6 Mos; Baseline, 12 Mos
Population: All participants who enrolled in the study and completed the scale at the designated time point.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Standard of Care
Number analyzed (Participants) | 56
units on a scale
  6 Mos: number analyzed (Participants) | 48
  6 Mos | 0.1 [0.0 to 0.2]
  12 Mos: number analyzed (Participants) | 33
  12 Mos | 0.1 [0.0 to 0.2]

ADVERSE EVENTS:
Arm/Group | Standard of Care
Serious Adverse Events (participants affected / at risk) | 1/56
Other Adverse Events (participants affected / at risk) | 10/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (N=56)
Oesophagitis (Gastrointestinal disorders) | 1 (1)
Dementia alzheimer's type (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (N=56)
Dementia alzheimer's type (Nervous system disorders) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days